CLINICAL TRIAL: NCT06952699
Title: A Randomized, Double-Blinded, Placebo-Controlled, Dose-Finding, Adaptive Trial to Evaluate the Safety, Tolerability, and Efficacy of TAK-360 in Participants With Narcolepsy Without Cataplexy (NT2)
Brief Title: A Study of TAK-360 in Adults With Narcolepsy Without Cataplexy (NT2)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-360-2001; 2024-517711-70-01 (EU CTIS Number)
Record Dates: First submitted 2025-04-23; First posted 2025-05-01 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Narcolepsy Type 2
Keywords: Narcolepsy without Cataplexy; NT2; TAK-360

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TAK-360 (Experimental): Participants will receive TAK-360 tablets, orally, for 4 weeks.
  Interventions: Drug: TAK-360
- Placebo (Placebo Comparator): Participants will receive TAK-360 matching-placebo tablets, orally, for 4 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: TAK-360 — TAK-360 tablet.
  Arms: TAK-360
Other: Placebo — TAK-360 matching placebo tablet.
  Arms: Placebo

SUMMARY:
Narcolepsy without cataplexy or Narcolepsy Type 2 (NT2) is a lifelong condition that makes people very sleepy during the day, regardless of how much sleep they get at night. People with NT2 may fall asleep suddenly, have trouble staying awake during the day, or may not be able to sleep well at night. They may have difficulty thinking clearly, paying attention, or remembering things, during the day. These symptoms can make daily activities like driving, working, or caring for their families challenging, impacting their quality of life. Orexin is a chemical made in the brain that helps keep a person awake and alert. TAK-360 acts like orexin. Previous studies have shown that medicines that act like orexin may keep people awake.

The main aim of this study is to learn how safe TAK-360 is and how well adults with NT2 tolerate it. Researchers also want to find out if TAK-360 can help people with NT2 stay awake and determine the right dosage needed to do that.

Participants will be randomly (by chance, like drawing names from a hat) assigned to get either TAK-360 or placebo in the treatment period. The placebo is a pill that looks just like TAK-360 but does not have any medicine in it. Using a placebo helps researchers learn about the real effect of the treatment.

ELIGIBILITY:
Key Inclusion Criteria:

1. The participant weighs greater than equal or to (≥)40 kilograms (kg) and has a body mass index (BMI) between 16 and 38 kilograms per meter square (kg/m^2) [inclusive].
2. The participant has a documented, current diagnosis of NT2.

Key Exclusion Criteria:

1. The participant has a current medical disorder associated with excessive daytime sleepiness (EDS) other than NT2.
2. The participant has medically significant thyroid disease.
3. The participant has a history of cancer in the past 5 years. (This exclusion does not apply to participants with carcinoma in situ [such as basal cell carcinoma] that has been treated and is stable, or who have been stable without further treatment. These participants may be included after approval by the medical monitor).
4. The participant has any of the following viral infections based on a positive test result: Hepatitis B surface antigen (at screening), hepatitis C virus (HCV) antibody (at screening), human immunodeficiency virus (HIV) antibody/antigen (at screening).
5. The participant has a clinically significant history of head injury or head trauma.
6. The participant has history of epilepsy, seizure, or convulsion (exception for a single febrile seizure in childhood).
7. The participant has a history of cerebral ischemia, transient ischemic attack (<5 years from screening), intracranial aneurysm, or arteriovenous malformation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2026-08-20 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With at Least One Treatment-emergent Adverse Event (TEAE) | Up to 15 Weeks
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product. A TEAE is defined as any event emerging or manifesting at or after the initiation of treatment with a study intervention or medicinal product or any existing event that worsens in either intensity or frequency following exposure to the study intervention or medicinal product.

SECONDARY OUTCOMES:
Change from Baseline at Week 4 in Epworth Sleepiness Scale (ESS) Total Score | Baseline, Week 4
  The ESS provides individuals with 8 different situations of daily life and asks them how likely they are to fall asleep in those situations (scored 0 to 3) and to try to imagine their likelihood of dozing even if they have not actually been in the identical situation; the scores are summed to give an overall score of 0 to 24. Higher scores indicate stronger subjective daytime sleepiness, and scores below 10 are considered to be within the normal range.
Change from Baseline at Week 4 in Mean Sleep Latency on the Maintenance of Wakefulness Test (MWT) | Baseline, Week 4
  The MWT evaluates a person's ability to remain awake under soporific conditions for a defined period of time. Because there is no biological measure of wakefulness, wakefulness is measured indirectly by the inability or delayed tendency to fall asleep. This tendency to fall asleep is measured via electroencephalography-derived sleep latency in the MWT. The MWT consists of four 40-minute sessions done 2 hours apart. Sleep latency in each session will be recorded. Participants will be required to stay awake in between the 4 sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (30):
- United States (12):
  - Takeda Site 14, Redwood City, California
  - Takeda Site 10, Santa Ana, California
  - Takeda Site 1, Colorado Springs, Colorado
  - Takeda Site 13, Brandon, Florida
  - Takeda Site 3, Orlando, Florida
  - Takeda Site 4, St Louis, Missouri
  - Takeda Site 8, Denver, North Carolina
  - Takeda Site 6, Huntersville, North Carolina
  - Takeda Site 5, Cincinnati, Ohio
  - Takeda Site 2, Columbia, South Carolina
  - Takeda Site 7, San Antonio, Texas
  - Takeda Site 11, Norfolk, Virginia
- China (3):
  - Takeda Site 28, Beijing, Beijing Municipality
  - Takeda Site 29, Guangzhou, Guangzhou
  - Takeda Site 27, Shanghai, Shanghai Municipality
- France (2):
  - Takeda Site 17, Montpellier, Hérault
  - Takeda Site 15, Paris
- Italy (3):
  - Takeda Site 22, Rome, Lazio
  - Takeda Site 31, Verona, Veneto
  - Takeda Site 23, Bologna
- Japan (6):
  - Takeda Site 24, Kohoku-ku, Yokohama-Shi, Kanagawa
  - Takeda Site 9, Kumamoto, Kumamoto
  - Takeda Site 30, Urasoe-Shi, Okinawa
  - Takeda Site 20, Shinjuku-ku, Tokyo
  - Takeda Site 26, Sumida-Ku, Tokyo
  - Takeda Site 12, Yodogawa-ku, Osaka-shi, Ôsaka
- South Korea (3):
  - Takeda Site 16, Junggu, Daegu Gwang'yeogsi
  - Takeda Site 19, Suwon, Gyeonggido
  - Takeda Site 21, Seoul, Seoul Teugbyeolsi
- Takeda Site 18, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/f4aacba8d8fb4c8f??page=1&idFilter=TAK-360-2001